CLINICAL TRIAL: NCT07031180
Title: The Effect of an Educational Intervention in Patient's Knowledge and Self-care Skills in Adult Patients With Venous Leg Ulcer in Outpatient Clinic of "Azienda ULSS 6 Euganea": a Two-arm, Single Centre Randomized Controlled Trial
Brief Title: Educational Interventions in Venous Leg Ulcer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Padova (Other)
Collaborators: Azienda Ulss 6 Euganea (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: VLU-2024-01
Record Dates: First submitted 2025-06-12; First posted 2025-06-22 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Venous Leg Ulcers
Keywords: venous leg ulcer; education; randomized controlled trial; knowledge; self-care skills
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): The video recordings will be made available to patients randomized to the experimental/intervention group by providing a QR code linked to the Youtube or other similar platform in order to be played by a digital device already available to patients and caregivers. It will be played for the first time at the end of the first study visit after all assessments have been completed. Patients and caregivers will be encouraged to play the video recordings as they need and prefer.
  Interventions: Other: educational video
- Control group (Active Comparator): The control group will not receive the additional educational video but will receive the standard of care and an educational pamphlet.
  Interventions: Other: educational pamphlet (standard educational intervention)

INTERVENTIONS:
Other: educational video — The experimental educational intervention will consist of professional video recordings that will cover the following topics:
  1. Disease knowledge (VLU)
  2. Medication management
  3. The importance of compression therapy
  4. Diet and physical activity The video recordings' contents will result from a review of the literature and guidelines, which will be later reviewed by a panel of experts in VLU. The video will be recorded by experienced video-maker and by a group of volunteers who will be the actors.
  Arms: Intervention group
Other: educational pamphlet (standard educational intervention) — The educational brochure is an educational intervention already in use at the setting involved in the study.
  Arms: Control group

SUMMARY:
Background: Venous ulcers are skin lesions caused by impaired blood circulation. In Western countries, about 1% of the population is affected, and approximately 3% those over 80 years old. Venous leg ulcers tend to become chronic; a lesion is defined as chronic when it does not progress towards spontaneous healing. The treatment of these lesions inevitably involves long healing times, which results in increased healthcare costs. Moreover, venous leg ulcers have recurrence rates ranging from 18% to 28%. For this reason, it is important to support patients affected by or at risk of venous ulcers during their healing process or for prevention.

Objectives: The primary objective of the study is to assess the superiority of the educational interventions to the standard therapeutic education, in improving the patient's/caregiver's self-efficacy, after 4 weeks, 3, 6 and 12 months from the educational intervention begin. The secondary objectives are to clinically assess the impact of the educational intervention in decreasing healing time and recurrence rates and in patients' well-being after 12 months of follow-up. Additionally, the Well-being of Wounds Inventory (WOW-I) questionnaire will be validated in its Italian version.

Methods: the study is a two arm moncentric randomized-controlled trial. The participants will be randomly assigned into two groups. The control group will receive an educational intervention through a pamphlet, which represents the standard education received in the outpatient clinics involved in the study. The intervention group instead will receive an experimental educational intervention through video played specifically for this study. The socio-demografic, health and ulcer related factors will be collected and the questionnaires: venous leg ulcer knowledge (VLUK), Venous Leg Ulcer Self-Efficacy Tool (VeLUSET) and Well-being Of Wounds Inventory (WOW I) will be administered to the patients during the outpatient clinic visit, before the treatment and after 4 weeks, 3 and 6 months after the intervention. The study also includes a telephonic follow up at 12 months from the start carried out to assess if the patient's venous ulcer has healed or recurred.

DETAILED DESCRIPTION:
Background:

Venous Leg Ulcers (VLU) are skin lesions occurring in the lower limbs stem from increased venous pressure, resulting in vessel dilation and fluid stagnation in the leg's lower regions. This condition is a complication of chronic venous insufficiency, damaging vessel walls and surrounding tissues. In Western countries, about 3 per cent of the population over 80 years old are affected.

In Italy, the prevalence of this disease is constantly increasing among adults, particularly the elderly, who often have concomitant diseases.

In clinical settings, treating VLU commonly encounters prolonged healing periods and recurrent occurrences, leading to escalated treatment expenses and patient discomfort. Patients report pain, sleep disturbances, wound smell, impaired mobility, altered body image, decreased vitality and disappointment with treatment leading to a physical, psychological, and social distress, markedly diminishing their perceived quality of life.

Due to the chronicity and prevalence of these ulcers, patients or their caregivers are often involved in VLU management and self-care. The last includes maintaining health, monitoring, and managing one's health condition. Maintenance is the phase in which the patient prevents injury or recurrence by acting on the reduction of risk factors, monitoring is the process of observing signs and symptoms, and finally management includes how the patient responds to the eventual signs and symptoms . It is known as a barrier to self-management of VLU to not receive adequate health information, this prevents the patient or family member to maintain health, monitor signs and symptoms and manage the injury.

It is very important to make the patient aware of their health condition, what the risk factors, complications, protective factors, and the types of treatment of signs and symptoms are. Non-invasive ulcer treatments encompass local dressings targeting lesion itself and adjacent skin, and compression therapy. Substantial evidence in literature proves compression therapy's efficacy in accelerating healing compared to sole local dressing application. Furthermore, a properly applied compression therapy reduces pain, pressure and volume overload in the venous system. Given the high recurrence rates at 12 months, from 18% to 28%, post-wound healing, continued preventive measures, particularly compression therapy, prove pivotal in mitigating relapse risk.

Unfortunately, many patients do not or only partially adhere to compression treatment. Adherence is influenced by people's beliefs about the usefulness of treatment and their awareness and knowledge of their disease. Increased knowledge about their disease improves patients' ability to involve themselves in self-care and leads them to avoid risk behaviour. To increase knowledge and prevent recurrences, educational interventions are needed to enable patients to fully understand the disease and to competently apply skin care and preventive therapy, promoting effective self-management. However, patient education consistency across different healthcare settings remains variable, with limited scientific evidence on intervention efficacy.

Educational interventions on VLU patients in outpatient's clinic lack clear guidelines about the method and is still operator dependent. If it is not always guaranteed through a standardized tool, it can be completely missing in case of high workload in the outpatient clinic as reported by clinicians involved in this care setting. According to the Baquerizo Nole study (2015), illustrative video recordings appear to be effective in improving patients' knowledge. However, this result is not statistically significant due to the small number of patients enrolled in previous studies.

Study design:

This study is a monocentric randomized controlled, open-label trial that involves a design with 2 parallel groups and a 1:1 allocation, to test the superiority of the experimental intervention in increasing the levels of knowledge and self-efficacy of patients with VLU versus standard of care. Patients will be randomised using block randomisation in order to prevent imbalance between the two groups.

A parallel longitudinal prospective sub study is dedicated to the validation of the Italian version of the Well-being Of Wounds Inventory questionnaire (WOW I).

The primary objective of the study is to assess the superiority of the educational interventions to the standard therapeutic education, in improving the patient's/caregiver's self-efficacy, after 4 weeks, 3, and 6 months from the educational intervention begin.

Moreover, as secondary objectives, the study aims to clinically assess the effect of the intervention on patient well-being throughout the follow-up period and, at the long-term, to determine the impact of the educational intervention on reducing healing time and recurrence rates after a 12-month follow-up period.

Furthermore, the enrolled patients will be asked to fill the Well-being Of Wounds Inventory (WOW I) questionnaire in order to validate it in its Italian version and collect valuable information about the well-being of the target population.

Setting and data collection methods:

The study will be conducted from the Italian clinical centres of the "Azienda ULSS 6 Euganea" in Veneto region.

The data will be collected in 14 months after IEC approval, probably starting in the autumn of 2024. Socio-health and demographic information will be gathered, and the patient will also be asked to complete the questionnaires 'Venous Leg Ulcer Knowledge (VLUK)' (Appendix 1), 'Venous Leg Ulcer Self Efficacy Tool (VeLUSET)' (Appendix 2), and "Well-being Of Wounds Inventory (WOW I)" (Appendix 3). The questionnaires will be collected using a company smartphone or tablet through the REDCap platform.

The data will be collected anonymously. During the patient's enrollment (clinic visit), the researcher will give to the patient a QR code, which the patient will use to complete the questionnaires for data collection.

Study duration:

The study will last one year after enrolment, three follow-ups are planned for the evaluation of primary outcomes. The first follow up will occur after 4 weeks ± 7 days (t2) after delivery of the educational video, the following follow ups will be after 3 months ± 7 days (t3) and 6 months ± 7 days (t4); if a patient will be healed before the conclusion of the follow ups this will exit the study and be classified as healed.

As for the secondary outcome of patient's well-being the investigator will assess it through the WOW I questionnaire during patient enrolment, later it will be reassessed 7±2 days (t1) after the first administration. Finally, 12 months (t5) after delivery of the educational video, there will be a long term follow up by telephone in which the patient will be asked when healing occurred (time) and if there were any recurrences (same lesion or other areas). Data collection forms will be available in the e-CRF.

Statistical analysis:

Descriptive analysis will summarize the baseline characteristics of the two randomized groups. Mean and standard deviation (if the assumption of and normality holds) or median and interquartile ranges will be provided for the analysis of continuous variables, proportions and frequency for categorical variables.

T-tests, paired sample t-tests, Wilcoxon Mann-Whitney, ANOVA for repeated measures, chi-square tests will be used when appropriate for comparison of continuous and categorical variables between the two groups or for comparison of variables in the same group pre- and post-treatment.

For analysis of survival, the Kaplan-Maier curve and log rank test will be used.

In case of imbalance between groups, multivariable generalized linear models will be used.

For the validation of the WOW I questionnaire will be conducted a parallel sub study with a longitudinal prospective non-interventional design. Analysis of data from the WOWI will be performed, regarding reproducibility, calculating intra-class correlations as an indicator of test-retest at enrolment and after one week) reliability; discriminant validity will be assessed by comparing the scores of respondents with poor, moderate, or good status as assessed by the VAS scale related to well-being in the EQ-5D; convergent validity will be established by comparing subscale scores with scores on the 'well-being' sub-scale of the Cardiff Wound Impact Schedule - CWIS.

All the analyses will be performed using R-4.3.3.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years;
* with venous leg ulcer;
* who understand Italian language;
* who is able to read and understand the questions;
* who attending to the nursing clinics involved in the study;
* who have given consent to participate in the study;
* who use a smart device with an internet connection or with caregiver able to provide the smart device as video player.

Exclusion Criteria:

* with cognitive impairment;
* who have an ankle-arm index/Winsor's index (ABI) less than 0.90. / with arterial insufficiency
* patients with arterial or mixed-origin ulcers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
The level of patient's knowledge | From enrollment to the end of treatment at 6 months
  A primary outcome of this study is the change of the level of patient's knowledge about him/her disease. This outcome will assess by the administration pre and post the educational intervention of the "Venous Leg Ulcer Knowledge (VLUK)" questionnaire in its Italian version, that comprises 15 multiple-choice questions. The tool has a minimum score of 0 and a maximum of 15 where higher scores mean a better knowledge about VLU.
The level of patient's self-care ability | From enrollment to the end of treatment at 6 months
  A primary outcome of this study is the change of the level of patient's self-care ability in the management of him/her disease. This outcome will assess by the administration, pre and post the educational intervention, of the "Venous Leg Ulcer Self Efficacy Tool (VeLUSET)". The tool comprises 30 itemswith a score from zero to ten (minimum score 0, maximum score 300), higer scores indicate more elevated perception of self-care ability.

SECONDARY OUTCOMES:
VLU recurrence | 12 months after enrolment
  A secondary outcome is the number of recurrences of VLU in the participants at 12 months.
healing time | From enrollment to the end of treatment at 6 months
  A secondary outcome is the number of patients cured during follow-up. This will be assessed using the PUSH 3.0 instrument score.
The well-being | From enrollment to the end of treatment at 6 months
  A secondary outcome is the change of well-being in patients with VLU. This outcome will assess by the administration pre and post the educational intervention of the "Well-being Of Wounds Inventory questionnaire (WOW I)", wich include 19 items with a five points likert scale, higer scores indicate better well-being.

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda ULSS 6 Euganea, Padua, PD, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Balestroni G, Bertolotti G. [EuroQol-5D (EQ-5D): an instrument for measuring quality of life]. Monaldi Arch Chest Dis. 2012 Sep;78(3):155-9. doi: 10.4081/monaldi.2012.121. Italian. PMID 23614330
- [Background] Baquerizo Nole KL, Yim E, Van Driessche F, Lamel SA, Richmond NA, Braun LR, Kirsner RS. Educational interventions in venous leg ulcer patients. Wound Repair Regen. 2015 Jan-Feb;23(1):137-40. doi: 10.1111/wrr.12247. Epub 2015 Feb 13. No abstract available. PMID 25487073
- [Background] Bobbink P, Pugliese MT, Larkin P, Probst S. Nurse-led patient education for persons suffering from a venous leg ulcer in outpatient's clinics and homecare settings: A scoping review. J Tissue Viability. 2020 Nov;29(4):297-309. doi: 10.1016/j.jtv.2020.08.006. Epub 2020 Aug 29. PMID 32907753
- [Background] Brown A. Evaluating the reasons underlying treatment nonadherence in VLU patients: introducing the VeLUSET Part 1 of 2. J Wound Care. 2014 Jan;23(1):37, 40, 42-4, passim. doi: 10.12968/jowc.2014.23.1.37. PMID 24406542
- [Background] Carradice D. Superficial venous insufficiency from the infernal to the endothermal. Ann R Coll Surg Engl. 2014 Jan;96(1):5-10. doi: 10.1308/003588414X13824511650498. PMID 24417822
- [Background] Huang Y, Hu J, Xie T, Jiang Z, Ding W, Mao B, Hou L. Effects of home-based chronic wound care training for patients and caregivers: A systematic review. Int Wound J. 2023 Nov;20(9):3802-3820. doi: 10.1111/iwj.14219. Epub 2023 Jun 5. PMID 37277908
- [Background] Kapp S, Miller C. The experience of self-management following venous leg ulcer healing. J Clin Nurs. 2015 May;24(9-10):1300-9. doi: 10.1111/jocn.12730. Epub 2014 Nov 24. PMID 25422075
- [Background] Martinato M, Ranzato C, Faggian E, Foletto M, Moreal C, Guidone N, Acar AS, Masiero F, Beghin F, Peruzzo S, Gregori D, Comoretto RI. Knowledge assessment among subjects with chronic venous leg ulcer in outpatient setting: Translation and adaptation of a tool to identify subjects at risk of poor understanding. Wound Repair Regen. 2023 Sep-Oct;31(5):679-687. doi: 10.1111/wrr.13107. Epub 2023 Jul 17. PMID 37368793
- [Background] O'Brien JA, Finlayson KJ, Kerr G, Edwards HE. Testing the effectiveness of a self-efficacy based exercise intervention for adults with venous leg ulcers: protocol of a randomised controlled trial. BMC Dermatol. 2014 Oct 3;14:16. doi: 10.1186/1471-5945-14-16. PMID 25277416
- [Background] Price P, Harding K. Cardiff Wound Impact Schedule: the development of a condition-specific questionnaire to assess health-related quality of life in patients with chronic wounds of the lower limb. Int Wound J. 2004 Apr;1(1):10-7. doi: 10.1111/j.1742-481x.2004.00007.x. PMID 16722893
- [Background] Protz K, Dissemond J, Seifert M, Hintner M, Temme B, Verheyen-Cronau I, Augustin M, Otten M. Education in people with venous leg ulcers based on a brochure about compression therapy: A quasi-randomised controlled trial. Int Wound J. 2019 Dec;16(6):1252-1262. doi: 10.1111/iwj.13172. Epub 2019 Aug 16. PMID 31418532
- [Background] Raffetto JD, Ligi D, Maniscalco R, Khalil RA, Mannello F. Why Venous Leg Ulcers Have Difficulty Healing: Overview on Pathophysiology, Clinical Consequences, and Treatment. J Clin Med. 2020 Dec 24;10(1):29. doi: 10.3390/jcm10010029. PMID 33374372
- [Background] Weller CD, Buchbinder R, Johnston RV. Interventions for helping people adhere to compression treatments for venous leg ulceration. Cochrane Database Syst Rev. 2016 Mar 2;3(3):CD008378. doi: 10.1002/14651858.CD008378.pub3. PMID 26932818
- [Background] Zulec M, Rotar Pavlic D, Zulec A. The Effect of an Educational Intervention on Self-Care in Patients with Venous Leg Ulcers-A Randomized Controlled Trial. Int J Environ Res Public Health. 2022 Apr 12;19(8):4657. doi: 10.3390/ijerph19084657. PMID 35457524